CLINICAL TRIAL: NCT06831305
Title: Bacterial Colonization of Nails With Methacrylic Coating in Relation to the Formation of Biofilms and Healthcare-associated Infections
Brief Title: Bacterial Colonization on Nails Covered With a Methacrylic Coating
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: 0120-301/2024-2711-3
Record Dates: First submitted 2025-01-31; First posted 2025-02-18 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-01

CONDITIONS: Bacterial Colonization
Keywords: methacrylates; nails; desinfection; transmission of infections

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- natural nails (Active Comparator): Alcohol hand sanitizer 3ml applied into hands, spread over hands up to the wrist and rubbed until dry on natural nails.
  Interventions: Diagnostic Test: Comparison of microbiological sampling on natural nails
- methaacrylic nails (Active Comparator): Alcohol hand sanitizer 3ml applied into hands, spread over hands up to the wrist and rubbed until dry on methaacrylic nails
  Interventions: Diagnostic Test: Comparison of microbiological sampling on methacrylic nails

INTERVENTIONS:
Diagnostic Test: Comparison of microbiological sampling on natural nails — Comparison of microbiological sampling before and after hand desinfection
  Other Names: natural nails
  Arms: natural nails
Diagnostic Test: Comparison of microbiological sampling on methacrylic nails — Comparison of microbiological sampling on methacrylic nails
  Arms: methaacrylic nails

SUMMARY:
In the research, the investigators will monitor the bacterial colonization of nails coated with a methacrylic coating

DETAILED DESCRIPTION:
It is known that the hand hygiene of healthcare workers is extremely important in order to prevent health-related infections. The effectiveness of hand disinfection can be affected by aspects of hand hygiene such as long nails and fingernail applications. In order to determine whether and to what extent fingernails applied among healthcare workers pose a risk of transmission of potentially pathogenic bacteria, and until what day artificial fingernails are safe in healthcare workers, the investigators will monitor bacterial colonization on nails with UV-cured methacrylic fingernails lamp and compared it with a control group of natural nails without application.

ELIGIBILITY:
Inclusion Criteria:

* nurses, doctors and respiratory physiotherapists employed in high-risk wards for patients
* healthy nail surface and cuticle

Exclusion Criteria:

* subjects with damaged nails or cuticles
* operating room staff using surgical hand brushing and staff in general nursing wards.

Ages: 16 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of microbial colonization between natural and methacrylate nails | From day 1st to the end of treatment on day 14th

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia